CLINICAL TRIAL: NCT05364489
Title: Efficacy, Safety and Exploratory Clinical Study of Bevacizumab Combined With Oxaliplatin and TAS-102 in First-line Treatment of Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hong Zong, Chief Physician，Department of Oncology, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOT-CRC-1LT
Record Dates: First submitted 2022-04-27; First posted 2022-05-06 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Advanced Colorectal Cancer
Keywords: CRC; Bevacizumab; Oxaliplatin; TAS-102; first-line treatment
MeSH Terms: interventions — Oxaliplatin; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab combined with Oxaliplatin and TAS-102 (Experimental): Efficacy, safety and exploratory clinical study of Bevacizumab combined with Oxaliplatin and TAS-102 in first-line treatment of advanced colorectal cancer
  Interventions: Drug: Bevacizumab combined with Oxaliplatin and TAS-102

INTERVENTIONS:
Drug: Bevacizumab combined with Oxaliplatin and TAS-102 — Bevacizumab (Anda, Qilu Pharmaceutical): 5 mg/kg, repeated every 2 weeks, administered by intravenous drip (ivgtt).
  Oxaliplatin: 85 mg/m2, repeated every 2 weeks, by intravenous infusion (ivgtt). TAS-102: 35 mg/m2 (maximum single dose 80 mg), orally, twice a day, on days 1 to 5, repeated every 2 weeks.
  Continuous administration until disease progression, death, toxicity intolerance, withdrawal of informed consent, or other reasons specified in the protocol; for patients who still benefit after comprehensive evaluation after initial disease progression, the investigator may decide whether to continue the treatment with the experimental drug .

SUMMARY:
This study is a single-arm, prospective, open-label observational clinical study to evaluate the efficacy and safety of Bevacizumab combined with Oxaliplatin and TAS-102 in patients with advanced unresectable rectal cancer.

DETAILED DESCRIPTION:
Eligible subjects received Bevacizumab in combination with Oxaliplatin and the TAS-102 investigational drug, and Bevacizumab and Oxaliplatin were administered intravenously on day 1 of each cycle. Medicine, every 14 days as a course of treatment, TAS-102 orally administered, 35mg/m2 (maximum single dose 80mg), bid, orally on the 1st to 5th days, 2 weeks as a course of treatment.

Patients were treated until objective disease progression, worsening symptoms, unacceptable toxicity, death, or withdrawal of consent, whichever occurred first. Clinicians will comprehensively evaluate according to clinical treatment guidelines and clinical practice treatment principles. For patients who still benefit after progression, the investigator can decide whether to continue the treatment with Bevacizumab combined with Oxaliplatin and TAS-102. Efficacy objectives were assessed after all subjects completed treatment/termination visits. Subjects were assessed for safety throughout the study period through laboratory tests and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

1. age: ≥18 years and ≤75 years;
2. ECOG score 0~1 points;
3. advanced colorectal cancer patients
4. According to RECIST1.1 criteria, there is at least one measurable target lesion, and tumor imaging evaluation is performed within 28 days before the first dose;
5. Expected survival time ≥ 12 weeks;
6. Major organ function is normal, that is, the following criteria are met:

（1）Routine blood examination standards must meet: ANC ≥1.5×109/L; PLT≥90×109/L; Hb ≥90g/L (no blood transfusion within 14 days); (2) Biochemical tests should meet the following criteria: ALB≥30g/L; (no ALB transfusion within 14 days); TBIL≤Upper limit of normal (ULN); ALT and AST≤2.5 times upper limit of normal (ULN), if liver metastasis , then ALT and AST≤5ULN; alkaline phosphatase≤2.5 times the upper limit of normal (ULN); BUN and Cr≤1.5×ULN and creatinine clearance rate≥50mL/min (CockcroftGault formula); (3) Cardiac ultrasound and echocardiography: left ventricular ejection fraction (LVEF≥55%); (4) QT interval (QTcF) corrected by Fridericia method of 18-lead ECG in females <470 ms; 7. For premenopausal or surgically sterilized female patients: Consent to abstinence or use of effective contraception during treatment and for at least 7 months after the last dose of study treatment; 8. Voluntarily joined the study and signed the informed consent.

Exclusion Criteria:

1. Patients who have received first-line standard therapy;
2. Previous antitumor therapy or radiation therapy for any malignant tumor;
3. concurrently receiving anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy, or immunotherapy;
4. Has undergone major surgical procedures not related to colorectal cancer within 4 weeks prior to enrollment, or the patient has not fully recovered from such surgical procedures;
5. Serious heart disease or discomfort, including but not limited to the following:

   * Diagnosed history of heart failure or systolic dysfunction (LVEF < 50%)
   * High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate >100 bpm, significant ventricular arrhythmia (eg, ventricular tachycardia), or higher-grade AV block (ie, Mobitz II second-degree AV block or third-degree AV blocklag)
   * Angina pectoris requiring antianginal drug treatment
   * Clinically significant heart valve disease
   * ECG showing transmural myocardial infarction
   * Poorly controlled hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg)
6. Inability to swallow, bowel obstruction, or other factors that interfere with drug taking and absorption;
7. Known history of allergies to the drug components of this regimen; history of immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
8. Pregnant or lactating female patients, female patients of childbearing potential with a positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period and within 7 months after the last study drug;
9. Serious comorbidities or other comorbidities that would interfere with planned treatment, or any other condition in which the patient is considered unsuitable for participation in this study by the investigator.

Dropout/Rejection Criteria:

1. The efficacy and/or safety evaluation cannot be performed due to the medication not prescribed in this protocol;
2. Participating in other anti-tumor treatments while participating in this study will be assessed by the investigator as affecting the efficacy evaluation.

Termination criteria:

1. The subject withdraws informed consent and requests to withdraw;
2. During the course of the study, the subject has a pregnancy event;
3. Subjects who cannot tolerate toxicity;
4. Disease progression;
5. Other circumstances in which the investigator considers it necessary to withdraw from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months
  Defined as the time from randomization to tumor progression in any aspect or death from any cause（Unit: month）. Assessed according to RECIST 1.1 criteria, analysis of this indicator included tumor evaluation results during study treatment and follow-up. If the patient has several indicators that can be determined as PD, the first indicator is used for PFS analysis; recurrence, new lesions or death are considered to have reached the study endpoint 1. The patient uses other systemic or targeted observation targets. Lesional anti-tumor therapy is also considered tumor progression.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 24 months
  Defined as the number of subjects whose tumors shrank or remained stable for a certain period of time, including complete remission (CR) and partial remission (PR), during the period from the time the subject received the treatment regimen of this study to the progression of the subject's disease in the analysis data set The percentage of the total population (unit: %).
  Evaluation method: Objective tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria). Subjects must have measurable tumor lesions at baseline. The efficacy evaluation criteria are divided into complete remission (CR), partial remission (PR), stable disease (SD), and progressive disease (PD) according to RECIST 1.1 criteria. Subjects assessed as CR, PR, and SD were confirmed after 3 weeks (at the next protocol-specified efficacy assessment).
Objective response rate (ORR) | Up to 24 months
  It is defined as the number of subjects with the best response effect as complete remission (CR) or partial remission (PR) during the period from the start of the subjects receiving the treatment regimen of this study to the progression of the subjects' disease in the total number of subjects in the analysis data set. percentage of the population（%）.
Overall survival (OS) | Up to 24 months
  Defined as the time from randomization to death from any cause（Unit: month）.
Drug-Related Safety Indicators | Up to 36 months
  Exposure to the investigational drug and incidence, nature, and severity of adverse events, including serious adverse events（n，%）。

IPD SHARING:
Plan to Share IPD: No